CLINICAL TRIAL: NCT04492800
Title: A Hair Loss Prevention Study for Patients With Advanced Pancreatic Cancer Utilizing Scalp Cooling
Brief Title: Hair Loss Prevention Study for Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HRI-ScalpCooling-001
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Paxman Scalp Cooling Device (Other): Patients will undergo scalp cooling via the Paxman Scalp Cooling device for the first 3 cycles of treatment. Cooling will consist of precooling (30 minutes); infusion cooling (will vary depending upon the length of time to infuse the chemotherapy) and post infusion cooling (90 minutes).
  Interventions: Device: Paxman Scalp Cooling Device

INTERVENTIONS:
Device: Paxman Scalp Cooling Device — Cooling will consist of precooling (30 minutes); infusion cooling (will vary depending upon the length of time to infuse the chemotherapy) and post infusion cooling (90 minutes).

SUMMARY:
Pilot study intended for hair loss prevention in patients with pancreatic cancer who are receiving treatment containing nab-paclitaxel, gemcitabine and cisplatin.

DETAILED DESCRIPTION:
Patients with pancreatic cancer who are receiving treatment containing nab-paclitaxel, gemcitabine and cisplatin will experience hair preservation with the use of the Paxman scalp cooling device, at the end of three, 3 week cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial
* >18 years of age on day of signing informed consent
* Diagnosis of pancreatic cancer and scheduled to receive treatment with a regimen containing nab-paclitaxel, gemcitabine and cisplatin

Exclusion Criteria:

* Grade 1 alopecia
* Existing history of scalp metastases or the presence of scalp metastases is suspected
* No history of previous cancers within the past 5 years
* CNS malignancies (either primary or metastatic)
* Cold sensitivity, cold agglutinin disease, cryoglobulinemia, cryofibrinogenemia, cold migraine, cold urticaria, post-traumatic cold dystrophy
* Imminent bone marrow ablation chemotherapy
* Imminent skull radiation
* Previously received or scheduled to undergo skull irradiation
* Severe liver or renal disease from any etiology as patient may not be able to metabolize or clear the metabolites of the chemotherapeutic agent
* Skin cancers including melanoma, squamous cell carcinoma and Merkel cell carcinoma
* Small cell carcinoma of the lung
* Solid tumors that have a high likelihood for metastasis in transit
* Squamous cell carcinoma of the lung

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hair Preservation | 28 to 84 days
  Patients will experience hair preservation defined as alopecia Grade 0 or 1 versus Grade 2 as defined by the CTCAE Version 5.0

SECONDARY OUTCOMES:
Patient Comfort | 1 to 84 days
  Patient's comfort while receiving scalp cooling using the Paxman scalp cooling device by asking one Likert scale question (comfortable or uncomfortable)
Chemotherapy-Induced Alopecia Distress | 1 to 84 days
  Identify chemotherapy-induced alopecia distress by utilizing the chemotherapy-induced alopecia distress scale (CADS) with scores ranging from 17-68 with a higher score indicating distress

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mirabella, PhD, RN, CHPN, Principal Investigator — HonorHealth Research Institute - Bisgrove
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States